CLINICAL TRIAL: NCT01457560
Title: Study to Assess the Immunogenicity and Reactogenicity of DTPa-HBV-IPV Mixed With Hib Vaccine in Healthy Infants, Followed by a Dose of the Same Vaccine Administered Simultaneously With One Dose of Oral Polio Vaccine (OPV)
Brief Title: Immunogenicity and Reactogenicity of DTPa-HBV-IPV/Hib Vaccine Followed by the Same Vaccine and Oral Polio Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 217744/060
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis B; Acellular Pertussis; Haemophilus Influenzae Type b; Diphtheria; Tetanus; Poliomyelitis
Keywords: Oral polio vaccine (OPV); DTPa-HBV-IPV/Hib vaccine
MeSH Terms: conditions — Hepatitis B; Haemophilus Infections; Diphtheria; Tetanus; Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: DTPa-HBV-IPV/Hib (Infanrix hexa™); Biological: OPV

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib (Infanrix hexa™) — Three doses administered intramuscularly
Biological: OPV — One dose administered orally

SUMMARY:
This study will assess the immunogenicity and safety of the GlaxoSmithKline (GSK) Biologicals' (formerly SmithKline Beecham Biologicals') combined DTPa-HBV-IPV/Hib (Infanrix hexa™) vaccine administered in the 3rd, 5th, 11th month of life. The last dose of DTPa-HBV-IPV/Hib will be given simultaneously with one dose of OPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be checked at study entry. If any of these criteria does not apply, the subject is not eligible for inclusion in the study.

* Healthy male and female subjects in the ≥12 and <16 weeks of life at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parents/guardians of the infant after they have been advised of the risks and benefits of the study in a language which they clearly understood, and before performance of any study procedure.

Exclusion Criteria:

The exclusion criteria will be checked at study entry and at each following visit. If any of these criteria applies at study entry, the subject is not eligible for inclusion in the study. If any of these criteria becomes applicable during the study, the subject should be withdrawn.

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of chronic immunosuppressants or other immune-modifying drugs within three months before vaccination).
* Administration of a vaccine not foreseen by the study within 30 days before each dose of the study vaccines and ending 30 days after.
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, polio and/or Hib disease.
* History of /or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio and/or Hib disease or infection.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of seizures or of any neurological disease at study entry.
* Administration of immunoglobulins and/or any blood products since birth, or planned administration during the study period.
* Acute disease at the time of enrolment.

Ages: 12 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2000-02; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to the components of the study vaccine in terms of number of subjects with antibody titres greater than or equal to cut off values | One month after the second dose and one month after the third dose of the primary vaccination course ( Month 3 and Month 9)

SECONDARY OUTCOMES:
Immunogenicity with respect to the components of the study vaccine in terms of number of subjects with antibody titres greater than or equal to cut off values | Before the first dose ( Month 0 )
Immunogenicity with respect to the components of the study vaccine in terms of antibody titers | Before the first dose (Month 0), one month after the second dose and one month after the third dose of the primary vaccination course ( Month 3 and Month 9).
Immunogenicity with respect to the components of the study vaccine in terms of number of subjects with vaccine response | One month after the second dose, and one month after the third dose of the primary vaccination course (Month 3 and Month 9).
Immunogenicity with respect to the components of the study vaccine in terms of antibody titres greater than or equal to cut off values | One month after the second dose, and one month after the third dose of the primary vaccination course (Month 3 and Month 9).
Number of subjects with solicited and unsolicited adverse events | After each dose of the study vaccines (Month 0, Month 3 and Month 9) and overall
Number of subjects with serious adverse events | During the study period (Month 0 to Month 9)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Van Der Meeren O, Kuriyakose S, Kolhe D, Hardt K. Immunogenicity of Infanrix hexa administered at 3, 5 and 11 months of age. Vaccine. 2012 Apr 5;30(17):2710-4. doi: 10.1016/j.vaccine.2012.02.024. Epub 2012 Feb 18. PMID 22349525
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 217744/060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 217744/060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 217744/060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 217744/060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register